CLINICAL TRIAL: NCT04834908
Title: A Prospective Randomized Multi-center Open Label Phase 1/2 Study to Evaluate the Safety and Efficacy of Equine COVID-19 Antiserum [F(ab')2](BSVEQAb) Plus Standard of Care in Comparison to Standard of Care Alone in COVID-19 RT-PCR Positive Patients
Brief Title: Evaluation of Equine Antibody Treatment in Patients With COVID 19 Infection
Acronym: PROTECT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed as no eligible patient.
Sponsor: Bharat Serums and Vaccines Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSV_EQ-AB_20_08
Record Dates: First submitted 2021-03-23; First posted 2021-04-08 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: SARS-CoV-2 Infection
Keywords: 2019 Novel Coronavirus Disease; COVID19; Coronavirus Disease 2019
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Clinical phase 1 and phase 2 studies have been planned to be conducted. The phase 1 study will be conducted on two dosages to find the safety and tolerability in patients. Each patient will receive either of the dose BSVEQAb - 5 mg/kg or 10 mg/kg body weight and all will receive standard of care
  Based on the results of phase 1 study the phase 2 shall be initiated. In phase 2 study one group will receive the tolerable dose of BSVEQAb selected along with standard of care. The second group will receive only standard of care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equine COVID-19 Antiserum [F(ab')2] (BSVEQAb) Along with Standard of care (Experimental): Dose of BSVEQAb - 5 mg/kg or 10 mg/kg body weight. It is administered as a single dose intravenously after diluting in 100 -150 ml saline. The infusion will be done over 1 to 2 hours.
  Standard of care for treatment of COVID-19 positive patients
  Interventions: Biological: Equine COVID-19 Antiserum; Drug: Standard of care
- Standard of care. (Active Comparator): Treatment as per current treatment guidelines and institutional practice for COVID-19 positive patients will be administered
  Interventions: Drug: Standard of care

INTERVENTIONS:
Biological: Equine COVID-19 Antiserum — Equine COVID-19 antiserum is a polyclonal antibody and it contains Equine COVID-19 immune globulin G.
  Other Names: F(ab)2, BSVEQAb, EqAb-COV-19
  Arms: Equine COVID-19 Antiserum [F(ab')2] (BSVEQAb) Along with Standard of care
Drug: Standard of care — Standard of care for COVID 19 infection based on the current guidelines and institutional practice will be provided

SUMMARY:
This is a Prospective, Randomized, Multi-center, Open label, Phase 1/2 study to Evaluate the Safety and Efficacy of Equine COVID-19 Antiserum [F(ab')2].

BSV has developed Equine COVID-19 antiserum from horse serum for the use in COVID-19 infection. The indication proposed is to provide passive immunization to the COVID-19 infected patient thereby reducing the viral load and prevention of disease progression.

Clinical phase 1 and phase 2 studies have been planned to be conducted. The phase 1 study will be conducted on two dosages to find the safety and tolerability in patients. Based on the results of phase 1 study the phase 2 shall be initiated.

ELIGIBILITY:
Inclusion Criteria:

1. Age Phase 1: ≥ 18 years to ≤ 55 years Phase 2: ≥ 18 years to ≤ 65 years
2. Are male or non-pregnant females who agree to contraceptive requirements.
3. Patients with RT-PCR confirmed COVID-19 in ≤ 72 hours prior to randomization [Ct ≥ 24].
4. Have SpO2<94% (range 90-93%) on room air.
5. Have one or more of the following- dyspnea, fever, cough, respiratory rate ≥ 24 per minute and heart rate up to 120 per minute.
6. Patients who agree to participate in the study and follow all study related procedures

Exclusion Criteria:

1. Require mechanical ventilation
2. Have oxygen saturation less than or equal to 89 percent
3. Patients re-infected with SARS-CoV-2
4. Suspected or proven serious active bacterial fungal viral or other infection
5. Patients with positive skin test with IP
6. Patients with known equine allergies or past medical history of serum sickness
7. Patient who are HIV, HCV, HbsAg positive or immunocompromised
8. Patients with significant co-morbidities at screening
9. Moribund state
10. Pregnant or nursing women
11. Participating in other clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Phase 1 Unexpected serious adverse events | Up to Day 28
  Number of patients with one or more unexpected serious adverse event(s) (SAEs) considered by the investigator to be related to study drug administration [Baseline through Day 28]
Phase 2 Patients turning COVID-19 negative (RT-PCR negative) | Day 5
  Proportion (percent) of patients turning COVID-19 negative
Phase 2 Patients turning COVID-19 negative (RT-PCR Negative) | Day 7
  Proportion (percent) of patients turning COVID-19 negative

SECONDARY OUTCOMES:
Phase 1 Patients turning COVID-19 negative (RT-PCR Negative) | Day 5
  Proportion (percent) of patients patients turning COVID-19 negative
Phase 1 Patients turning COVID-19 negative (RT-PCR Negative) | Day 7
  Proportion (percent) of patients patients turning COVID-19 negative
Phase 1 Exploratory outcome | Day 10
  Proportion (percent) of patients turning COVID-19 negative (RT-PCR negative)
Phase 1 Exploratory outcome | Day 14
  Proportion (percent) of patients turning COVID-19 negative (RT-PCR negative)
Phase 1-Exploratory outcome | Day 3 from Baseline
  Mean reduction in WHO clinical progression scale
Phase 1-Exploratory outcome | Day 5 from Baseline
  Mean reduction in WHO clinical progression scale
Phase 1- Exploratory outcome | Day 7 from Baseline
  Mean reduction in WHO clinical progression scale
Phase 1- Exploratory outcome | Day 14 from Baseline
  Mean reduction in WHO clinical progression scale
Phase 1- Exploratory outcome | Day 28 from Baseline
  Mean reduction in WHO clinical progression scale
Phase 2 Unexpected serious adverse events | up to Day 28
  Number of patients with one or more unexpected serious adverse event(s) (SAEs) considered by the investigator to be related to study drug administration
Phase 2 Patients turning COVID-19 negative (RT-PCR negative) | Day 10
  Proportion (percent) of patients turning COVID-19 negative
Phase 2 Patients turning COVID-19 negative (RT-PCR negative) | Day 14
  Proportion (percent) of patients turning COVID-19 negative
Phase 2 Change in WHO clinical progression scale | Day 3 from baseline
  Mean reduction in WHO clinical progression scale
Phase 2 Change in WHO clinical progression scale | Day 5 from baseline
  Mean reduction in WHO clinical progression scale
Phase 2 Change in WHO clinical progression scale | Day 7 from baseline
  Mean reduction in WHO clinical progression scale
Phase 2 Change in WHO clinical progression scale | Day 14 from baseline
  Mean reduction in WHO clinical progression scale
Phase 2 Change in WHO clinical progression scale | Day 28 from baseline
  Mean reduction in WHO clinical progression scale

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Jagannathan, Principal Investigator — Bharat Serums and Vaccines Ltd
Locations (1):
- Jehangir Hospital, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No